CLINICAL TRIAL: NCT04157036
Title: Comparative Evaluation of Preoperative Methylprednisolone or Ibuprofen on Anesthetic Efficacy of Inferior Alveolar Nerve Blocks in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Evaluation of Methylprednisolone or Ibuprofen on Efficacy of Nerve Blocks With Symptomatic Irreversible Pulpitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID halted recruitment for 2 years. A majority of patients eligible for the study had already taken preoperative analgesics, which disqualified them for the study.
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Neal, Director, Advanced Specialty Program in Endodontics, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRNMMC-2019-0249
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2020-02

CONDITIONS: Irreversible Pulpitis
Keywords: Inferior alveolar nerve block; Symptomatic irreversible pulpitis; Preoperative steroid; Preoperative NSAID
MeSH Terms: interventions — Ibuprofen; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 800mg Ibuprofen (Experimental): Subject will take 800mg of Ibuprofen 45 minutes prior to anesthetic delivery.
  Interventions: Drug: Ibuprofen
- 40mg Methylprednisolone (Experimental): Subject will take 40mg of Methylprednisolone 45 minutes prior to anesthetic delivery.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ibuprofen — Subject will take 800mg Ibuprofen 45 minutes prior to anesthetic delivery
  Arms: 800mg Ibuprofen
Drug: Methylprednisolone — Subject will take 40mg Methylprednisolone 45 minutes prior to anesthetic delivery
  Arms: 40mg Methylprednisolone

SUMMARY:
This prospective, randomized, double-blind study will compare the effect of oral premedication of ibuprofen and methylprednisolone on the anesthetic efficacy of an Inferior Alveolar Nerve Block (IANB) in adult patients with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
The NPDS Endodontic clinic is a referral base clinic. All scheduled and/or emergency (sick-call) patients undergo a thorough clinical and radiographic examination. Patients will be asked to enroll in this prospective study when a diagnosis of symptomatic irreversible pulpitis is established, nonsurgical root canal treatment is indicated and they meet all study inclusion/exclusion criteria. An investigator, not involved in treatment, will explain the study and answer all question(s). Those that agree to participate will be consented and enrolled.

To qualify for this study, each patient had a tooth that fulfilled the criteria for a clinical diagnosis of symptomatic irreversible pulpitis: a vital mandibular posterior tooth actively experiencing pain; a prolonged response to cold testing using Green Endo-Ice (1,1,1,2 tetrafluoroethane; Hygenic Corp, Akron, OH) and had not taken any analgesics within the past 8 hours.

Exclusion criteria are as follows: any person under the age of 18 years; allergies or sensitivities to Ibuprofen or Methylprednisolone; allergies or sensitivities to local anesthetics or sulfites; were pregnant or nursing; medical condiditons that contraindicate the ingestion of Ibuprofen or Methylprednisolone, such as : active or latent peptic ulcers, Crohn's Disease, ulcerative colitis, gastroesophageal refulx, systemic fungal infections, active herpetic infections, asthma, open-angle glaucoma, osteoporosis or cirrohsis; has as a medical condition requiring the use of steroid medications; or had a history of a serious medical condition preventing routine dental treatment. Patients with no response to cold testing, presence of periradicular pathology (other than a widened periodontal ligament), or the lack of vital coronal pulpal tissue upon endodontic access were also excluded from the study. Thus, confirming the clinical diagnosis of irreversible pulpitis.

After written informed consent is obtained, a study subject will rate their pain prior to administration of an analgesic on a visual analogue scale (VAS) (14). The VAS used is 10 cm in length and divided into four categories. No pain defined at 0 mm, mild pain 1mm to 50mm, moderate pain 51mm to 74mm, and severe pain is defined as 75mm or greater. Subjects' will rate their pain on this scale at specific timeframes during treatment dependent upon when anesthetic success is achieved.

Two oral medications are compared in this study: 800mg Ibuprofen and 40mg Methylprednisolone. The medications are blinded to the subject and the provider. Each medication will be compounded, visibly identical and labeled as either A or B by the Investigational Pharmacy Department at WRNNMC (the PI will be provided the code in a sealed envelope). A third party, not involved in the study, will distribute the blinded medication to the provider for administration to the subject. Forty-five minutes after oral administration of the blinded medication, an inferior alveolar nerve block (IANB) and long buccal nerve block (LBNB) will be administered to each subject. Prior to the injection, the anesthetic injection site is dried with a 2 x 2 gauze, then 20% benzocaine topical anesthetic gel is placed at the site for 1 minute using a cotton tip applicator. Standard IANB and LBNB injections are administered with a 27-gauge, 1 ¼ in. needle attached to an aspirating syringe. Each cartridge of anesthetic used contains 34mg of 2% lidocaine with 0.017mg of epinephrine. Each subject receives 2 full cartridges of anesthetic in total with 1.5 cartridges given as an IANB and 0.5 cartridges given as a LBNB. Each cartridge was measured in millimeters from the end of the aluminum cap to the stopper. This distance was found to be 50mm in length, therefore at the 25mm mark on every cartridge a line was drawn dividing all the anesthetic solution into halves. All injections were administered by one of three board certified endodontic staff members.

After anesthetic delivery, the subject will remain in a semi-supine position for fifteen minutes. The subject is questioned for lip numbness in five-minute intervals for up to fifteen minutes. If the subject does not achieve lip numbness, the nerve block is considered missed, patient care will continue with additional anesthesia administered. Data collection will not occur afterward. A missed block is different than a failed block. A failed block hit the target area, however due to the inflammatory nature of the disease process, the patient still is not completely anesthetized and requires additional anesthesia. Our study is trying to suppress that inflammatory process with the steroid medication, therefore hopefully leading to more successful blocks. A missed block does not hit the target area and therefore the patient does not exhibit signs of anesthesia, therefore the effect the medication has on that block is irrelevant at that point and cannot be measured because additional anesthesia is needed to begin the procedure. The subject becomes a patient and his or her participation in the study is ended. Non-surgical root canal treatment will be completed following the NPDS Endodontic Dept. Standard of Care for that particular tooth. The following methodology will be followed for the remaining enrolled subjects. It should be noted all of the following procedures normally would be Standard of Care for patients presenting for Endodontic treatment at NPDS. The consenting of subjects, prescribing of either of the oral medications, and recording of VHS scores, during and shortly after the Endodontic procedure, are the research components of this study.

If after the fifteen minutes (60 minutes after the administration of ibuprofen or methylprednisolone) lip numbness is perceived, teeth are isolated with a rubber dam and endodontic access is initiated. These subjects will complete the entire study. Subjects are informed to raise a hand to alert the dental team if they feel pain during the endodontic procedure. The goal of treatment is a thorough pulpal debridement of each canal without pain during the procedure. If pain occurs, the procedure is immediately stopped and the subject rates their pain on a VAS scale. The success of the IANB is defined as the ability to access and instrument the canal(s) without pain (VAS score of 0) or mild pain (VAS score of 1 -50mm).

Rubber dam isolation is removed for those who rated their pain as moderate or severe during access preparation. A supplemental buccal infiltration injection is administered in the alveolar mucosa near the apex (apices) buccal to the tooth under treatment utilizing a 27-gauge short needle and a cartridge of 68mg 4% articaine with 0.017mg epinephrine. All injections are given by one of three board certified endodontic staff members. Rubber dam isolation is reapplied five minutes after the supplemental injection and endodontic access is continued. The supplemental buccal injection is considered a success if endodontic access, initial file placement and canal debridement is completed without pain (VAS score of 0) or mild pain (VAS score of 1-50mm). Once again, if the subject indicates pain during access or instrumentation, the procedure is stopped and the subject rates their pain on a VAS scale. If pain is moderate (VAS score of 51-75mm) or severe (VAS score of 76-100) the supplemental buccal infiltration injection will be recorded as a failure (the subject will remain in the study) and an intraosseous injection is given as described by previous authors (15, 16). Rubber dam isolation is reapplied five minutes after the intraosseous injection and endodontic access is continued. Following the same protocol as with the supplemental buccal injection, if the subject indicates pain during access or instrumentation, the procedure is stopped and the subject rates their pain on a VAS scale. All injections were administered by one of three board certified endodontic staff members. As a last resort, if pain still occurs after the intraosseous injection, an intrapulpal injection is given and no VAS scores will obtained after the intrapulpal injection.

Obturation of the root canal (completion of treatment) may or may not be accomplished in one appointment. A thorough pulpal debridement is acceptable and the subject will be scheduled to complete treatment. Regardless of how many appointments it takes to complete the root canal, subjects will be finished with the study once they turn in the completed pain journal (following the first appointment).

After treatment is completed, each subject is given a pain journal and asked to note their pain six, twelve, twenty-four and forty-eight hours after treatment. The journal is returned to the provider at the follow up appointment for completion of root canal therapy. Following enrollment of the last subject, the code will be revealed and the data analyzed.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Has a vital mandibular posterior tooth experiencing pain
* Has a prolonged response to thermal cold testing using Green Endo Ice (1, 1, 1, 2 tetraflouroethane
* Diagnosis of symptomatic irreversible pulpitis

Exclusion Criteria:

* Has taken an analgesic within the past 8 hours
* Allergies or sensitivities to Ibuprofen or Methylprednisolone
* Allergies or sensitivities to local anesthetics or sulfites
* Pregnant or nursing
* Has a history of a serious medical condition preventing routine dental treatment
* Has a medical condition requiring the use of steroid medications
* Active or latent peptic ulcers
* Crohn's Disease
* Ulcerative colitis
* Gastroesophageal reflux
* Systemic fungal infection
* Active herpetic infection
* Asthma
* Open-angle glaucoma
* Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Analgesic Effect on Nerve Block | 48 hours
  To compare the effect of two oral pre-medications, ibuprofen and methylprednisolone, on the anesthetic efficacy of the inferior alveolar nerve block (IANB) using a VAS scale in patients with symptomatic irreversible pulpitis. The scale is 100mm long. If the subject experiences pain during the procedure, he/she will mark the scale. If it is marked at 50mm or lower, the nerve block is considered a success (no or mild pain), if it is marked above 50mm, the nerve block failed and supplemental anesthetic will be administered. We will be looking at whether the preoperative medications had an effect on the nerve block success.

SECONDARY OUTCOMES:
Analgesic Effect on Supplemental Anesthesia Techniques | 48 hours
  If the subject reports pain during the procedure, a supplemental injection will be administered. Our secondary objective is to compare the efficacy of a supplemental injection of 4% articaine with 1:100,000 epinephrine, if administered, using a VAS scale, in the two experimental groups. The scale is 100mm long. If the subject experiences pain after supplemental anesthesia has been administered, he/she will again mark the scale. If it is marked at 50mm or lower, the supplemental anesthesia is considered a success (no or mild pain), if it is marked above 50mm, the anesthesia failed and more supplemental anesthetic will be administered. We will be looking at whether the preoperative medications had an effect on the supplemental anesthesia success.
Analgesic Effect on Post-Operative Pain | 48 hours
  At the conclusion of treatment we will be asking the subjects to complete a pain diary for the following 48 hours. Our tertiary objective is to compare the level of postoperative pain, using a VAS scale, in both experimental groups, to include whether supplemental injections were needed or not. The scale is 100mm long. There are three categories of pain: mild pain (1-50mm), moderate pain (51-75mm) and severe pain (76-100mm). We will be accessing on whether the preoperative medications had an effect on postoperative pain based on these three categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share our data with any other Researchers.

REFERENCES:
- [Result] Nagendrababu V, Pulikkotil SJ, Veettil SK, Teerawattanapong N, Setzer FC. Effect of Nonsteroidal Anti-inflammatory Drug as an Oral Premedication on the Anesthetic Success of Inferior Alveolar Nerve Block in Treatment of Irreversible Pulpitis: A Systematic Review with Meta-analysis and Trial Sequential Analysis. J Endod. 2018 Jun;44(6):914-922.e2. doi: 10.1016/j.joen.2018.02.017. Epub 2018 Apr 27. PMID 29709297
- [Result] Aggarwal V, Singla M, Kabi D. Comparative evaluation of effect of preoperative oral medication of ibuprofen and ketorolac on anesthetic efficacy of inferior alveolar nerve block with lidocaine in patients with irreversible pulpitis: a prospective, double-blind, randomized clinical trial. J Endod. 2010 Mar;36(3):375-8. doi: 10.1016/j.joen.2009.11.010. PMID 20171350
- [Result] Fowler S, Drum M, Reader A, Beck M. Anesthetic Success of an Inferior Alveolar Nerve Block and Supplemental Articaine Buccal Infiltration for Molars and Premolars in Patients with Symptomatic Irreversible Pulpitis. J Endod. 2016 Mar;42(3):390-2. doi: 10.1016/j.joen.2015.12.025. Epub 2016 Jan 28. PMID 26831048
- [Result] Fowler S, Reader A, Beck M. Incidence of missed inferior alveolar nerve blocks in vital asymptomatic subjects and in patients with symptomatic irreversible pulpitis. J Endod. 2015 May;41(5):637-9. doi: 10.1016/j.joen.2015.01.029. Epub 2015 Mar 11. PMID 25770038
- [Result] Drum M, Reader A, Nusstein J, Fowler S. Successful pulpal anesthesia for symptomatic irreversible pulpitis. J Am Dent Assoc. 2017 Apr;148(4):267-271. doi: 10.1016/j.adaj.2017.01.002. Epub 2017 Feb 9. PMID 28190451
- [Result] Henry MA, Hargreaves KM. Peripheral mechanisms of odontogenic pain. Dent Clin North Am. 2007 Jan;51(1):19-44, v. doi: 10.1016/j.cden.2006.09.007. PMID 17185058
- [Result] Nagori SA, Jose A, Roy ID, Chattopadhyay PK, Roychoudhury A. Does methylprednisolone improve postoperative outcomes after mandibular third molar surgery? A systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2019 Jun;48(6):787-800. doi: 10.1016/j.ijom.2018.09.005. Epub 2018 Oct 9. PMID 30314709
- [Result] Collins SL, Moore RA, McQuay HJ. The visual analogue pain intensity scale: what is moderate pain in millimetres? Pain. 1997 Aug;72(1-2):95-7. doi: 10.1016/s0304-3959(97)00005-5. PMID 9272792
- [Result] Nusstein J, Reader A, Nist R, Beck M, Meyers WJ. Anesthetic efficacy of the supplemental intraosseous injection of 2% lidocaine with 1:100,000 epinephrine in irreversible pulpitis. J Endod. 1998 Jul;24(7):487-91. doi: 10.1016/S0099-2399(98)80053-8. PMID 9693577
- [Result] Reisman D, Reader A, Nist R, Beck M, Weaver J. Anesthetic efficacy of the supplemental intraosseous injection of 3% mepivacaine in irreversible pulpitis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1997 Dec;84(6):676-82. doi: 10.1016/s1079-2104(97)90372-3. PMID 9431539

DOCUMENTS (1):
  • Informed Consent Form (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT04157036/ICF_000.pdf